CLINICAL TRIAL: NCT03966755
Title: Unsaturated Fatty Acids to Improve Cardiorespiratory Fitness in Patients With Obesity and Heart Failure With Preserved Ejection Fraction: The UFA-Preserved2 Study
Brief Title: Unsaturated Fatty Acids to Improve Cardiorespiratory Fitness in Obesity and HFpEF
Acronym: UFA-Preserved2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM20016253
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Heart Failure With Normal Ejection Fraction
Keywords: Obesity; Heart failure with Normal Ejection Fraction; HFpEF; unsaturated fatty acids; cardiorespiratory fitness; dietary intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UFA dietary recommendations (Experimental): Dietary intervention aimed at increasing UFA consumption.
  Interventions: Behavioral: UFA dietary recommendations
- Standard dietary recommendations (No Intervention): Standard of care dietary recommendations as currently performed in the clinic (2015-2020 United States Department of Agriculture (USDA) Dietary Guidelines for Americans)

INTERVENTIONS:
Behavioral: UFA dietary recommendations — The face-to-face intervention will be performed by a research nutritionist that reviews the dietary recall and provides a list of commonly available foods rich in unsaturated fatty acids (UFA) (monounsaturated fatty acids (MUFA) and polyunsaturated fatty acids (PUFA)), together with individual instructions on how to integrate the recommended foods in the daily dietary pattern based on the dietary recall, and also to emphasize that the recommended food should be consumed as listed, and not as part of processed food (i.e., guacamole for avocado, hazelnut chocolate for nuts, pesto for olive oil, fish sticks for fatty fish). Extra-virgin olive oil or canola oil or nuts will be considered first choice for daily consumption of UFA-rich food, but a list of daily food substitutes will be also provided .
  Arms: UFA dietary recommendations

SUMMARY:
This study is designed to evaluate the effects of a diet rich in unsaturated fatty acids (UFA)-also known as 'healthy fats'-in patients with obesity and heart failure with preserved ejection fraction (HFpEF) on dietary consumption of UFA as well as fatty acids plasma levels.

DETAILED DESCRIPTION:
The study will evaluate participant's food consumption during 2 different 12-week periods. During one of the 12-week periods, participants will receive specific counseling and instructions on how to increase the consumption of food rich in healthy fats; during the other 12-week period they will receive general dietary recommendations following the Dietary Guidelines for Americans. There will be a 6-week break (washout) between the 12-week periods for a total of study period of 30 weeks. During each 12-week periods, the study will measure the effects of these dietary recommendations on dietary consumption and the fatty acids in their blood (primary endpoints).

ELIGIBILITY:
Major Inclusion Criteria:

* Body Mass Index (BMI) ≥30 kg/m2 (obesity) or total body fat percentage >25% in men and >35% in women
* A confirmed clinical diagnosis of stable HF (New York Heart Association (NYHA) class II-III) on maximally tolerated heart failure (HF) optimal medical regimen (without major changes in the prior month)
* Left Ventricular Ejection Fraction (LVEF)>50% documented in the prior 12 months

Major Exclusion Criteria:

* Concomitant conditions or treatment which would affect completion or interpretation of the study (i.e.,physical inability to walk or run on treadmill);
* Significant ischemic heart disease, angina, uncontrolled arterial hypertension, atrial fibrillation, moderate to severe valvular disease, chronic pulmonary disease, anemia (Hemoglobin<10 g/dL)
* Electrocardiography (ECG) changes (ischemia or arrhythmias) that limit maximum exertion during cardiopulmonary exercise test
* Comorbidity limiting survival
* Stage IV-V kidney disease (estimated Glomerular Filtration Rate<30)
* Fluid overload
* Pregnancy
* Current use of unsaturated fatty acids (UFA) supplement (i.e., omega-3).
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour dietary recall | At baseline, at 12 weeks, at 18 weeks, and at 30 weeks
  Measured with validated 24-hour dietary recall (non-self administered)
Change in dietary compliance (biomarkers) | At baseline, at 12 weeks, at 18 weeks, and at 30 weeks
  Measured by changes in biomarkers of unsaturated fatty acid consumption

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Carbone, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03966755/ICF_000.pdf